CLINICAL TRIAL: NCT05562778
Title: Evaluation of a Chatbot to Maximize Hereditary Cancer Genetic Risk Assessment in an Underserved Gynecology Population
Brief Title: Chatbot to Maximize Hereditary Cancer Genetic Risk Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-11024123
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Gynecologic Cancer; Hereditary Cancer Syndrome
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Intervention Model Description: 2-arm randomized controlled trial of a chatbot for personal/family history intake vs. usual care (intake via the clinician interview). Enrolled patients will be randomized in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chatbot (Experimental): Subjects will receive a text message initiating a chatbot conversation that relies on natural language processing to gather personal and family cancer. Subjects are identified by the chatbot as meeting National Comprehensive Cancer Network (NCCN) high-risk criteria. Next, subjects undergo pre-test genetic counseling via the chatbot and then clinicians are notified (via the chatbot portal) that the subject meets high-risk criteria. For subjects meeting high-risk criteria (based on the chatbot evaluation), the clinician will complete genetic counseling and recommend genetic testing during the visit. For subjects interested in genetic testing, the clinician will order genetic testing.
  Interventions: Other: Chatbot
- Usual Care (No Intervention): Personal and family cancer history will be collected by the clinician during the subject's visit. Clinicians will evaluate the patient's personal/family history according to National Comprehensive Cancer Network (NCCN) high-risk criteria. For subjects recognized by the clinician as meeting NCCN criteria, the clinician will complete genetic counseling and recommend genetic testing. For subjects interested in genetic testing, the clinician will order genetic testing.

INTERVENTIONS:
Other: Chatbot — A chatbot is a software program designed to simulate human conversation, typically via text. Chatbots utilize natural language processing to gather patient data, anticipate questions, and predict responses. In this study, the Chatbot will simulate a text-like conversation with patients via a smartphone and use this platform to deal with the time-consuming nature of family history collection. The chatbots can then triage the collected family history against medical guidelines to determine which patients warrant genetic testing. For those patients meeting criteria for genetic testing, the chatbot can offer pre-test education and assist physicians with ordering genetic testing for interested patients meeting high-risk criteria.
  Arms: Chatbot

SUMMARY:
In this study, the investigators aim to compare a mobile health platform, known as a 'chatbot,' that leverages artificial intelligence and natural language processing to scale communication, to 'usual care' that patients would receive. This comparison will enable the investigators to determine if the chatbot system can improve rates of recommendation for genetic testing among patients at elevated risk of harboring a familial cancer syndrome in an all-Medicaid gynecology clinic. Furthermore, the investigators aim to evaluate facilitators of inequity in regard to patient access to and utilization of genetic testing services.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older.
* Scheduled for a New Patient appointment in the gynecology clinic. Speaks and reads in English.
* Access to a telephone with texting capacity.
* Has not had prior genetic testing for hereditary cancer syndromes.

Exclusion Criteria:

* Under 18 years of age
* Has had previous genetic testing for hereditary cancer syndromes
* Does not read/speak in English
* Does not have access to a phone with texting capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion recommended genetic testing | 2 years
  The proportion of high-risk patients that are recommended genetic testing for familial cancer syndromes in the chatbot vs. usual care arms.

SECONDARY OUTCOMES:
Proportion completed recommended genetic testing | 2 years
  The proportion of high-risk patients who complete recommended genetic testing for familial cancer syndromes in the chatbot vs. usual care arms.
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, education, affordability, and social determinants of health. The validated survey known as the Hospital Anxiety and Depression Scale (HADS) will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the HADS survey has 7 questions each to assess depression and anxiety subscales. Scoring for each item ranges from 0 to 3, with 3 denoting highest anxiety or depression level, and 0 denoting the lowest. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, education, affordability, and social determinants of health. The validated survey known as the NCCN Distress Thermometer will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the NCCN Distress Thermometer allows patients to self report how much distress they have been experiencing in the past week on a scale from 0 (no distress) to 10 (extreme distress).
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, affordability, and social determinants of health. The validated survey known as the Satisfaction with genetic assessment will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the Satisfaction with genetic assessment includes the review of a patient's personal and family history with regards to cancer that was performed by the medical provider during the patient's Gynecology New Patient Visit. This is scaled from strongly agree to strongly disagree.
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, affordability, and social determinants of health. The validated survey known as the Satisfaction with Decision Scale will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the Satisfaction with Decision Scale will assess a patient's satisfaction with their decision to undergo genetic testing using 6 statements that a patient must agree or disagree with, scaled from strongly agree to strongly disagree.
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, affordability, and social determinants of health. The validated survey known as the Feelings about Genomic Testing Results (FACToR) survey Scale will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the Feelings about Genomic Testing Results (FACToR) survey asks 12 questions regarding how the patient felt after they received their genetic results, indicating within the past week if they had the specific feeling: not at all, a little, somewhat, a good deal, or a great deal.
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, affordability, and social determinants of health. The validated survey known as the Perceptions of Uncertainties in Genomic Sequencing (PUGS) survey will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the Perceptions of Uncertainties in Genomic Sequencing (PUGS) survey assesses patient's certainty about 8 aspects of their genetic testing, from 1 (very uncertain) to 5 (very certain).
Facilitator of inequity in the utilization of genetic services | 2 years
  The specific facilitators of inequity that affect the utilization of genetic testing services, among high-risk patients who decline recommended genetic testing. Examples of these facilitators include patient race, ethnicity, affordability, and social determinants of health. The validated survey known as the Patient Reported Utility (PrU) survey will enable these patients to identify various facilitators that influenced their decision not to complete genetic testing. Specifically, the Patient Reported Utility (PrU) that assesses how useful patients found certain outcomes of their test results, ranking from 1 (not at all useful) to 7 (extremely useful).
Barriers to genetic testing | 2 years
  The barriers (as identified through qualitative interviews) to genetic testing among high-risk patients who decline recommended genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa K Frey, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - NYP Brooklyn Methodist Hospital, Brooklyn, New York
  - NYP Lower Manhattan Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York
  - NYP Medical Group Queens, Queens, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bull LE, Webster EM, McDougale A, Howard D, Ahsan MD, Levi S, Grant B, Chandler I, Christos P, Sharaf RN, Frey MK. Protocol for Health Risk Information Technology-Assisted Genetic Evaluation (HeRITAGE): a randomised controlled trial of digital genetic cancer risk assessment in a diverse underserved gynaecology clinic. BMJ Open. 2024 Sep 5;14(9):e082658. doi: 10.1136/bmjopen-2023-082658. PMID 39237276